CLINICAL TRIAL: NCT07207187
Title: An Ambispective Efficacy Evaluation of the Karma Fixation System
Brief Title: Karma Ambispective Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Spinal Elements (Industry)
Collaborators: The Spine Network (Unknown)
Responsible Party: Sponsor
Other Study IDs: TSN-2025-SEK
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Subjects Treated With Karma Fixation System as Part of Their Spine Surgery
Keywords: Degenerative spine; Karma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Subjects treated with the Karma Fixation System as part of their spine surgery.: Subjects implanted with the Karma Fixation System in the lumbar spine as part of their spine surgery.

SUMMARY:
The purpose of this observational, multi-center, ambispective study is collect real world patient outcomes that characterize the effectiveness of the Karma Fixation System in the lumbar spine.

DETAILED DESCRIPTION:
This is a multicenter, observational, ambispective study of up to 100 patients across a maximum of 10 US sites. Retrospective data collection will be performed from preoperative up to the single prospective visit. Prospective data collection will include a one-time visit to obtain post-operative imaging. In the event a subject has a complete 12-month data set available retrospectively, the prospective visit may not be required.

PRIMARY ENDPOINTS:

- Fusion status at a minimum of 12-months postoperative (≥10 months post surgery)

SECONDARY ENDPOINTS:

* Procedure-or device-related serious adverse events (SAE)
* Patient reported outcomes if available included, Oswestry Disability Index (ODI), Back and leg pain as measured by Visual Analog Scale (VAS), 12-Item Short Form Health Survey (SF-12)

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature and age ≥ 18 years of age at the time of surgery
* Previously treated with the Karma Fixation System
* Has at least 12-months post-surgery imaging obtained including a minimum 2 view x-rays (lateral flexion and lateral extension) and CT scan, or willing to return to obtain imaging
* Be willing and able to comply with the study protocol requirements
* Be willing to sign the study-specific Informed Consent Document

Exclusion Criteria:

* Previous fusion or total disc replacement at the index level(s)
* Active systemic infection at the index level at the time of surgery
* Current active or suspected malignancy, or a cancer diagnosis that was ongoing during the patient's treatment and healing period
* Diagnosis of osteomalacia or Paget's bone disease
* Currently enrolled in a competing research study
* Currently incarcerated \
* Currently pregnant or plans to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will include a maximum of 10 US sites.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Fusion | 12 month post surgery (≥10 months post surgery)
  Fusion at treated levels as measured by x-rays and CT scan.

SECONDARY OUTCOMES:
Serious Adverse Events | Surgery through study completion
  Incidence of serious adverse events (SAE).
Change in Pain | Baseline and 12 months post surgery
  Pain improvement as measured by Visual Analog Scale (VAS), 0-100mm. Higher score indicates increased pain.
Change in Disability | Baseline and 12 months post surgery
  Disability improvement as measured by Oswestry Disability Index (ODI), 0-100%. High score indicates increase disability
Change in Quality of Life | Baseline and 12 months post surgery
  Improvement in qualify of life as measured by 12-item Short Form Health Survey (SF-12), 0-100. High score indicates increase quality of life.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Sonoran Spine, Gilbert, Arizona
  - Ascension St. Vincent's, Jacksonville, Florida
  - The Spine Institute of Louisiana, Shreveport, Louisiana
  - Neuroscience Specialist, Oklahoma City, Oklahoma